CLINICAL TRIAL: NCT04322357
Title: Impact and Interplay of Corticosteroid Regimen and Exercise Training on DMD Muscle Function
Brief Title: Twice Weekly Steroids and Exercise as Therapy for DMD
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB201901339; MD 180023 (Other Grant/Funding Number: U.S. Army Medical Research and Development Command); OCR27142 (Other: UF OnCore)
Record Dates: First submitted 2020-03-24; First posted 2020-03-26 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Duchenne Muscular Dystrophy (DMD)
Keywords: steroid side effects, low dose steroid regimen, exercise training therapy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — Prednisone; Glucocorticoids; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Daily Glucocorticoid (GC) (No Intervention): Existing data from age-matched, ambulatory, on daily GC therapy, and similar exclusion criteria will be selected from the ImagingDMD database to serve as a historical control.
- Twice weekly glucocorticoid with or without exercise (Active Comparator): Patients will be randomized to one of 2 groups:
  * Twice weekly prednisone alone for 12 months
  * Twice weekly prednisone for 6 months followed by twice weekly prednisone plus 6 months of structured, supervised and home-based exercise training.
  Interventions: Drug: Prednisone
- Daily glucocorticoid with exercise (Active Comparator): Patients on daily glucocorticoids will undergo 6 months of structured, supervised and home-based exercise training.
  Interventions: Drug: Prednisone; Behavioral: In-home Exercise Training; Drug: Prednisone plus exercise

INTERVENTIONS:
Drug: Prednisone — A 12-month treatment period with twice weekly, low-dose prednisone (dose of 0.75 mg/kg per day).
  Other Names: Glucocorticoid (GC)
  Arms: Daily glucocorticoid with exercise; Twice weekly glucocorticoid with or without exercise
Behavioral: In-home Exercise Training — For boys on current standard of care (daily glucocorticoid use), 6-months in-home, remotely supervised exercise training program involving a combination of aerobic and isometric leg strength exercises.
  Arms: Daily glucocorticoid with exercise
Drug: Prednisone plus exercise — Twice weekly prednisone for 6 months followed by twice weekly prednisone plus exercise for 6 months.
  Arms: Daily glucocorticoid with exercise

SUMMARY:
The study team will determine the potential of low dose twice weekly prednisone and whether exercise training can synergize to delay disease progression and improve muscle strength/physical function in boys with Duchenne muscular dystrophy (DMD). Current standard of care (daily prednisone) is associated with adverse side effects. Evidence from DMD mouse models suggest that weekly dosing provides same efficacy without side effects. Appropriate exercise may also benefit but this area has not been adequately explored.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of DMD confirmed by 1) clinical history with features before the age of five, 2) physical examination, 3) elevated serum creatine kinase level and 4) absence of dystrophin expression, as determined by immunostain or Western blot (<2%) and/or DNA confirmation of dystrophin mutation.
* Age 5.0 to 9 years: a lower age limit of 5.0 years is selected as children younger than that are likely unable to cooperate and comply with all of the exercise measures as needed. An upper age limit of 9 years has been set as boys with DMD tend to reach a rapid progression into a late ambulatory phase soon after this age.
* Ambulatory at the time of the first visit, defined as the ability to walk for at least 100 m without an external assistive device and able to climb four stairs.
* Aim 1 only: GC-naïve at baseline (and prior 6 months)
* Aim 2 only: on stable daily GC regimen for 6 months prior to baseline

Exclusion Criteria:

* Contraindication to an MR examination (e.g. aneurysm clip, severe claustrophobia, magnetic implants)
* Presence of unstable medical problems, significant concomitant illness including cardiomyopathy or cardiac conduction abnormalities
* Presence of a secondary condition that impacts muscle function or muscle metabolism (e.g. myasthenia gravis, endocrine disorder, mitochondrial disease)
* Presence of a secondary condition leading to developmental delay or impaired motor control (e.g. cerebral palsy)
* Presence of an unstable medical condition (e.g. uncontrolled seizure disorder)
* Behavioral problems causing an inability to cooperate during testing or understand exercise instruction
* Participation in other forms of drug or gene therapy during the period of the study

Ages: 5 Years to 9 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 89 (Estimated)
Dates: Start 2020-07-30 (Actual); Primary Completion 2025-09-05 (Estimated); Study Completion 2025-10-07 (Estimated)

PRIMARY OUTCOMES:
Change in BMI | Baseline up to 12 months
  Participant body mass index change (weight and height will be combined to report BMI in kg/m^2) over the course of one year

CONTACTS AND LOCATIONS:
Overall Officials: Tanja Taivassalo, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No